CLINICAL TRIAL: NCT03152890
Title: Insulin Therapy for Postreperfusion Hyperglycemia in Liver Transplantation
Brief Title: Insulin Therapy for Postreperfusion Hyperglycemia
Acronym: INS_LTPL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Prof, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Insulin_LTPL
Record Dates: First submitted 2017-05-03; First posted 2017-05-15 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hyperglycaemia (Diabetic); Liver Transplantation
Keywords: Insulin; Liver transplantation; Hyperglycemia
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: The study group receives a linear mixed effects model-proposed dose of insulin when hyperglycemia is noticed after reperfusion of liver graft.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The study group receives a linear mixed effects model-proposed dose of insulin when hyperglycemia is noticed after reperfusion of liver graft.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — If blood glucose level after reperfusion of liver graft exceeds 180 mg/dL, the insulin dose proposed by the linear mixed effects analysis is given as a bolus.

SUMMARY:
Glycemic control during liver transplantation is challenging especially after reperfusion of the liver graft. Insulin dose to treat postreperfusion hyperglycemia is retrospectively analyzed using historical data. The proposed dose then is prospectively applied to the patients to assess the adequacy of the insulin dose.

DETAILED DESCRIPTION:
Hyperglycemia is common during liver transplantation ,especially after graft reperfusion. Response to insulin is frequently unpredictable during postreperfusion period with no consensus or guidelines on glycemic control. The primary aim of this mixed retrospective/prospective study is to investigate the optimal insulin dose to treat hyperglycemia during the postreperfusion period of liver transplantation.

In the retrospective study, adult liver recipients (>18 years old) who underwent liver transplantation between 2004 and 2016 are reviewed. Delta glucose is the primary outcome variable defined as the difference in blood glucose levels before and after insulin administration. The relationship between the insulin dose and delta glucose is analyzed with a linear mixed effects analysis to find the optimal insulin dose to treat postreperfusion hyperglycemia.

In the prospective trial, the proposed insulin dose is administered to the patient who showed hyperglycemia after graft reperfusion. The frequency and magnitude of glucose reduction is the primary outcome. The secondary outcome is the incidence and degree of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Liver recipients who showed hyperglycemia (blood glucose >180mg/dL) after reperfusion of liver graft.

Exclusion Criteria:

* pediatric patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of blood glucose level 20 minutes after insulin administration | 20 minutes after insulin administration
  Insulin is administered immediately after baseline hyperglycemia (blood glucose >180 mg/dL) has been observed.
  Change of blood glucose level after insulin administration is calculated as (baseline glucose - glucose after insulin administration).

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No